CLINICAL TRIAL: NCT00115817
Title: The Effects of Atorvastatin on the Rho/Rho Kinase Pathway in Patients With Atherosclerosis
Brief Title: The Effects of Atorvastatin in Patients With Atherosclerosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: 2005P-000416
Record Dates: First submitted 2005-06-26; First posted 2005-06-27 (Estimated); Last update posted 2007-04-24 (Estimated); Status verified 2007-04

CONDITIONS: Atherosclerosis
MeSH Terms: conditions — Atherosclerosis | interventions — Atorvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Atorvastatin

SUMMARY:
The purpose of the study is to evaluate the effects of Atorvastatin.

The investigators want to find out if atorvastatin has other helpful qualities. The investigators are interested in finding out if medicines like atorvastatin are useful even in people who do not have high levels of bad cholesterol and would like to understand other mechanisms by which this medicine helps prevent further blood vessel disease.

Hypotheses:

1. Atorvastatin reduces Rho kinase activity (in leukocytes) rapidly, within days, in patients with atherosclerosis.
2. Any decrease in Rho kinase activity with statin therapy will be accompanied by improvement in familiar markers of atherosclerosis.

DETAILED DESCRIPTION:
The total study period is approximately 14 + 28 days. There will be a total of 5 visits: a screening visit, followed by visits at 0, 7, 14 and 28 days. (These dates may vary by approximately 2 days in the event of a weekend or holiday). At the baseline visit (day 0), patients will be randomly assigned to atorvastatin 10 mg/day (given as 1 placebo pill + 1 10mg pill), 80 mg/day (given as 2 40mg pills) or placebo (given as 2 placebo pills). Subjects will be asked to take 2 pills every day at the same time between 7 p.m. and 8 p.m., and record in a calendar/diary any side effects, missed doses, change in concomitant medication, or any other pertinent information. At each visit, blood will be collected for the following tests: 1) Lipid profile, 2) C-Reactive protein, 3) Rho kinase expression and activity in leukocytes, 4) nitric oxide synthase (NOS) expression/activity in platelets, and 5) leukocyte/monocyte adhesion/migration assays. Blood for hepatic and muscle tests (ALT, GGT and CK) to monitor for side effects will be determined at baseline and at 28 days and as clinically indicated. At each visit, patients will be questioned about compliance with study medication and any side effects. All patients will be encouraged to adhere to the NCEP-ATPIII recommended therapeutic life style. Subjects will be asked to resume any statin medications they were taking prior to enrollment upon completion of the study.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects aged 21 to 80 years
* Modified NCEP ATPIII guideline criteria should be met to initiate statin therapy
* Known stable atherosclerotic disease (diagnosed coronary, peripheral or carotid vascular disease) and/or diabetes mellitus (a coronary heart disease equivalent)
* Written informed consent with prior primary care physician approval

Exclusion Criteria:

* Inability to give consent
* Pregnancy
* Inability to withdraw statin therapy for a 6 week period
* Prior history of intolerance to statins
* Hepatic dysfunction (ALT or GGT > 2 times the upper limit of normal
* Elevated muscle enzymes (CK > 3 times the upper limit of normal)
* History of myopathy or myositis
* Evidence of active inflammatory, infectious or neoplastic disease
* Use of cyclosporine, fibric acid derivatives, nicotinic acid, erythromycin, azole antifungals, prednisone or any immunosuppressant
* Coronary artery bypass graft surgery or percutaneous coronary intervention within the preceding 3 months
* Acute coronary syndrome or myocardial infarction within the preceding 3 months
* History of life-threatening arrhythmias without an implantable cardioverter defibrillator
* Severe chronic congestive heart failure
* Severe anemia
* Serum creatinine > 3 mg/dl

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36
Dates: Start 2005-06; Study Completion 2007-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Selwyn, MD, Principal Investigator — Brigham and Womens Hospital
Locations (1):
- Brigham and Womens Hospital, Boston, Massachusetts, United States